CLINICAL TRIAL: NCT00735436
Title: Phase II Trial for Patients With Glioblastoma Multiforme (GBM) Treated With Gliadel Followed by Avastin Plus Irinotecan
Brief Title: A Study of Gliadel Followed by Avastin + Irinotecan for Glioblastoma Multiforme (GBM)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study enrollment was halted due to slow accrual.
Sponsor: Duke University (Other)
Collaborators: Eisai Inc. (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006308
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2012-12

CONDITIONS: Malignant Glioma; Glioblastoma Multiforme; Gliosarcoma
Keywords: Malignant glioma; Glioblastoma multiforme; GBM; Gliosarcoma; Gliadel; Carmustine; Irinotecan; CPT-11; Camptosar; Avastin; Bevacizumab
MeSH Terms: conditions — Glioma; Glioblastoma; Gliosarcoma | interventions — carmustine, poliferprosan 20 drug combination; Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gliadel/Avastin/CPT-11 (Other): Gliadel/Avastin/CPT-11
  Interventions: Drug: Gliadel/Avastin/CPT-11

INTERVENTIONS:
Drug: Gliadel/Avastin/CPT-11
  Other Names: bevacizumab; irinotecan

SUMMARY:
The primary objective of the study is to use 24 week survival to assess the efficacy of the combination of Gliadel followed by Avastin and irinotecan in the treatment of grade IV malignant glioma patients following surgical resection. The secondary objectives are to determine the progression-free survival following the combination of Gliadel followed by Avastin and irinotecan and to describe the toxicity of Gliadel followed by Avastin and irinotecan.

DETAILED DESCRIPTION:
This is a phase II study of the combination of Gliadel followed by Avastin and irinotecan in grade IV malignant glioma patients. The study will have survival and toxicity endpoints. Subjects will be identified by the investigator as those patients who have histologically documented grade IV malignant glioma (glioblastoma multiforme or gliosarcoma) with recurrent or progressive disease who are able to undergo a gross total resection (GTR).

Part I: Gliadel wafer- 1-8 wafers inserted at time of gross total resection. Treatment cycle is 42 days in length. For patients with ≥ Grade 1 toxicity will allow 84 days prior to beginning therapy with Avastin and Irinotecan (CPT-11).

Part II: Avastin Plus Irinotecan (Cycles 1-12) consists of the following (cycle length is 6 weeks):

* Irinotecan 125 mg/m2 (not taking enzyme-inducing anti-epileptic drugs (EIAEDs)) or 340 mg/m2 (taking EIAEDs) given every two weeks on days 1, 15, 29, etc.;
* If the patient has the uridine diphosphate (UDP) glucuronosyltransferase 1 family, polypeptide A1 (UGT1A1) polymorphism (7/7), they do not metabolize the irinotecan normally, so these patients will start out at a two dose level reduction; For patients on an EIAED, the starting dose will be 275 mg/M2, and for patients not on an EIAED, the starting dose will be 75 mg/M2;
* Avastin 10 mg/kg immediately after the irinotecan given every 2 weeks on days 1, 15, 29, etc.

The primary objective of this phase II study is to determine whether the administration of Gliadel wafers followed by Avastin and irinotecan to patients with recurrent GBM is a treatment regimen worthy of further investigation in a randomized clinical trial. The basis for making this decision will be the proportion of patients who survive at least 24 weeks after initiation of protocol treatment.

In the initial Phase I and II clinical trials, four potential Avastin-associated safety signals were identified: hypertension, proteinuria, thromboembolic events, and hemorrhage. The two major toxicities associated with irinotecan are myelosuppression and diarrhea. Side effects associated with Gliadel are seizures, brain edema (swelling), healing abnormalities, wound infection and body pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of WHO grade IV primary malignant glioma (glioblastoma multiforme or gliosarcoma). Patients have to be able to undergo a GTR.
* Age > or = 18 years
* Evidence of a unilateral, single focus of measurable central nervous system (CNS) neoplasm on contrast-enhanced MRI, unless medically contraindicated (CT scan will then be used)
* Patients must have < or = 2 disease progressions
* An interval of at least 4 weeks from the end of prior radiotherapy or one week from the end of a cycle of chemotherapy and enrollment on this protocol
* Karnofsky > or = 70%
* Hemoglobin > or = 9.0 g/dl, absolute neutrophil count (ANC) > or = 1,500 cells/microliters, platelets > or = 125,000 cells/microliters
* Serum creatinine < or = 1.5 mg/dl, serum glutamic-oxaloacetic transaminase (SGOT) and bilirubin < or = 1.5 times upper limit of normal
* Patients on corticosteroids must have been on a stable dose for 1 week prior to entry, if clinically possible, and the dose should not be escalated over entry dose level
* If patient received chemotherapy or investigational agent as part of their prior therapy, the patient must recover from all toxicities (> or = Grade 1) prior to enrollment on this protocol
* Signed informed consent approved by the Institutional Review Board
* No evidence of CNS hemorrhage on the baseline MRI or CT scans
* If sexually active, patients will take contraceptive measures for the duration of treatment as stated in the informed consent

Exclusion Criteria:

* Pregnancy or breast feeding. Women of childbearing potential must have a negative serum pregnancy test within 72 hours prior to treatment administration
* Multifocal disease
* Prior treatment with Gliadel
* Prior treatment with CPT-11 or Avastin
* Prior stereotactic radiosurgery or brachytherapy
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids
* Active infection requiring IV antibiotics
* Acute or chronic renal insufficiency (a glomerular filtration rate (GFR) <30 mL/min/1.73m2) or acute renal insufficiency of any severity due to hepato-renal syndrome or in the peri-operative liver transplantation period
* Inability, in the opinion of the study investigator, to comply with study and/or follow-up procedures
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored Avastin cancer study
* Life expectancy of less than 12 weeks
* Active malignancy, other than superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix within last five years
* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to Day 1
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis (> or = 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula, gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria at screening as demonstrated by urinalysis (urine protein)
* Known hypersensitivity to any component of Avastin
* Pregnancy (positive pregnancy test) or lactation. Use of effective means of contraception (men and women) in subjects of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-12; Primary Completion 2011-07 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, FRCPC, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- See also: Duke University Medical Center Clinical Trials — http://www.dukehealth.org/clinicaltrials
- See also: The Preston Robert Tisch Brain Tumor Center — http://www.cancer.duke.edu/btc

RESULTS

PARTICIPANT FLOW:
Groups:
- Gliadel/Avastin/CPT-11: Gliadel wafers (1-8) inserted at time of gross total resection. CPT-11 (Irinotecan): 125 mg/m2 (no enzyme-inducing anticonvulsant drugs) or 340 mg/m2 (enzyme-inducing anticonvulsant drugs) given every two weeks on days 1, 15, 29 of each 42 day cycle, up to 12 cycles. If the patient has the uridine diphosphate (UDP) glucuronosyltransferase 1 family, polypeptide A1 (UGT1A1) polymorphism (7/7), they do not metabolize the irinotecan normally, so these patients will start out at a two dose level reduction. For patients on an enzyme-inducing anti-epileptic drugs (EIAED), the starting dose will be 275 mg/M2, and for patients not on an EIAED, the starting dose will be 75 mg/M2. Avastin: 10 mg/kg immediately after the irinotecan given every 2 weeks on days 1, 15, 29 of each 42 day cycle.
Period: Overall Study
Arm/Group | Gliadel/Avastin/CPT-11
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gliadel/Avastin/CPT-11
Number analyzed (Participants) | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 55.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: 24-week Overall Survival
Description: The percentage of participants surviving 24 weeks from the start of study treatment
Time Frame: 24 weeks
Population: intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gliadel/Avastin/CPT-11
Number analyzed (Participants) | 18
percentage of participants | 77.8 [51.1 to 91.0]

2. Secondary Outcome: 24-week Progression-free Survival (PFS)
Description: The percentage of participants surviving 24 weeks from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of the first documented progression according to modified Macdonald criteria, or to death due to any cause.
Time Frame: 24 weeks
Population: intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gliadel/Avastin/CPT-11
Number analyzed (Participants) | 18
percentage of participants | 61.1 [35.3 to 79.2]

3. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Time in months from the start of study treatment to the date of first progression according to modified Macdonald criteria, or to death due to any cause. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve.
Time Frame: Time in months from the start of study treatment to the date of first progression according to modified Macdonald criteria or to death due to any cause, assessed up to 47 months
Population: intent-to-treat
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Gliadel/Avastin/CPT-11: Gliadel wafers (1-8) inserted at time of gross total resection. CPT-11 (Irinotecan): 125 mg/m2 (no enzyme-inducing anticonvulsant drugs) or 340 mg/m2 (enzyme-inducing anticonvulsant drugs) given every two weeks on days 1, 15, 29 of each 42 day cycle, up to 12 cycles. If the patient has the UGT 1A1 polymorphism (7/7), they do not metabolize the irinotecan normally, so these patients will start out at a two dose level reduction. For patients on an EIAED, the starting dose will be 275 mg/M2, and for patients not on an EIAED, the starting dose will be 75 mg/M2. Avastin: 10 mg/kg immediately after the irinotecan given every 2 weeks on days 1, 15, 29 of each 42 day cycle.
Arm/Group | Gliadel/Avastin/CPT-11
Number analyzed (Participants) | 18
months | 8 [3.2 to 15.8]

4. Secondary Outcome: Median Overall Survival (OS)
Description: Time in months from the start of study treatment to date of death due to any cause. Patients alive at last follow-up are censored as of that follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: Time in months from the start of study treatment to date of death due to any cause, assessed up to 47 months
Population: intent-to-treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gliadel/Avastin/CPT-11
Number analyzed (Participants) | 18
months | 13.5 [6.0 to 19.5]

5. Secondary Outcome: Incidence and Severity of Central Nervous System (CNS) Hemorrhage
Description: Incidence and severity of CNS hemorrhage
Time Frame: 47 months
Population: intent-to-treat
Measure: Number; unit: participants
Arm/Group | Gliadel/Avastin/CPT-11
Number analyzed (Participants) | 18
participants
  Grade 5 CNS Hemorrhage | 1
  Grade 4 CNS Hemorrhage | 0

6. Secondary Outcome: Incidence of Grade ≥ 4 Hematologic and ≥ Grade 3 Non-hematologic Toxicities
Description: Incidence of grade ≥ 4 hematologic and ≥ grade 3 non-hematologic toxicities
Time Frame: 47 months
Population: intent-to-treat
Measure: Number; unit: participants
Arm/Group | Gliadel/Avastin/CPT-11
Number analyzed (Participants) | 18
participants
  Grade >= 4 Hematologic Toxicity | 0
  Grade >= 3 Non-hematologic Toxicity | 2

ADVERSE EVENTS:
Time Frame: 47 months
Description: Adverse Events were collected for the study using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, but were converted to CTCAE version 4.0 for entry in ClinicalTrials.gov.
Arm/Group | Gliadel/Avastin/CPT-11
Serious Adverse Events (participants affected / at risk) | 8/18
Other Adverse Events (participants affected / at risk) | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gliadel/Avastin/CPT-11 (N=18)
Lung infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 3
Wound dihiscence (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Cognitive disturbance (Nervous system disorders) | 2
Encephalopathy (Nervous system disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Ischemia cerebrovascular (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gliadel/Avastin/CPT-11 (N=18)
Anemia (Blood and lymphatic system disorders) | 8
Eye disorders-Other, specify: decreased vision (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 1
Bronchial infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Wound infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Investigations-Other, specify: Ammonia elevated (Investigations) | 1
Investigations-Other, specify: Total Protein Elevated Intermittently (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 5
White blood cell decreased (Investigations) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Ataxia (Nervous system disorders) | 3
Cerebrospinal fluid leakage (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysphasia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Seizure (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Thromboembolic event (Vascular disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No